CLINICAL TRIAL: NCT06202924
Title: The Effect of Attention Focus on Muscle Strength and Balance in Individuals With Joint Hypermobility
Brief Title: Muscle Strength and Balance in Individuals With Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ali ZORLULAR, principal investigator, Gazi University
Other Study IDs: Joint Hypermobility
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-01

CONDITIONS: Joint Hypermobility; Balance; Muscle Strength
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Muscle Strength and Balance Assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Static balance assessment — Biodex stabilometer device will be used to evaluate the static balance of the participants.
Behavioral: Dynamic balance assessment: — Individuals' dynamic balance performances were evaluated with the Y balance test. Y balance test is a test method with proven validity and reliability in athletes and healthy subjects. (Intra-class correlation 0.99-1, Inter-class correlation 0.85-0.91).
Behavioral: Isokinetic strength evaluation: — Quadriceps muscle strength of the participants will be evaluated with an isokinetic dynamometer. Isokinetic dynamometers are considered the gold standard in muscle strength measurements. These devices have the ability to objectively report the amount of force produced by individuals at predetermined angular speed and joint range of motion.

SUMMARY:
Joint hypermobility is a clinical condition characterized by joints having a range of motion beyond their normal limits. Joint hypermobility (JH) makes the joints more vulnerable to trauma in individuals with increased joint range of motion, changes in neuromuscular reflexes and decreased joint position sense. Individuals with JH have difficulty in stabilization and end of extension range of motion compared to healthy individuals. Accordingly, findings such as balance problems and an increased risk of falling occur in these patients. Recent evidence suggests that children and adults with JH may be identified with seemingly unrelated, common clinical problems such as chronic fatigue, anxiety, and a range of gastrointestinal functional disorders.

The use of internal and external focus in learning motor skills is important in terms of performance and activity. In the external focus of attention (EF), attention is directed to movement and an environmental stimulus. In the internal focus (IF), attention is directed directly to body movements. In revealing positive effects in external focus; Methods such as metaphor, analogy, imaginary objects, mental analogies can be used. Adopting an external focus of attention (focusing on the effects of movements on the object or environment), as opposed to an internal focus of attention (focusing on body movements), has been found to significantly improve performance on a variety of tasks. For example, to improve balance performance, while a patient performs a single-leg balance task on a Bosu ball, the therapist may instruct the patient using an internal focus of attention such as "minimize movement of the feet." However, instructions can also be given externally by changing just one word, such as "minimize Bosu's movement." Additionally, a metaphor (e.g., "stand still as if stuck to Velcro"), analogy ("imagine being on top of a mountain, stay on the mountain!"), an object attached to the body ("keep the tape stuck to the chest still"), or the target of the movement An imaginary object (e.g., straight line) of which a mental image is obtained has been used within external focus instructions.

DETAILED DESCRIPTION:
Joint hypermobility is a clinical condition characterized by joints having a range of motion beyond their normal limits. Joint hypermobility (JH) makes the joints more vulnerable to trauma in individuals with increased joint range of motion, changes in neuromuscular reflexes and decreased joint position sense. Individuals with (external focus) EF have difficulty in stabilization and end of extension range of motion compared to healthy individuals. Accordingly, findings such as balance problems and an increased risk of falling occur in these patients. Recent evidence suggests that children and adults with JH may be identified with seemingly unrelated, common clinical problems such as chronic fatigue, anxiety, and a range of gastrointestinal functional disorders.

The benefit of an external focus of attention compared to an internal focus of attention to enhance motor skill learning and performance has been consistently demonstrated by a large body of evidence across different populations, tasks, and skill levels . These developments included tasks such as balance, running, agility performance, direction changing performance, force production, horizontal and vertical jumping performance. In general, an external focus of attention has been shown to produce more accurate performance, improved reaction time, and more efficient movement (e.g., reduced muscle activity). According to the constrained action hypothesis, an IF encourages broader involvement of cognitive processes due to greater reliance on conscious control strategies. These strategies interfere with the normal automatic control processes of the motor system. An EF, on the other hand, encourages these automatic control processes, thus further enhancing motor learning. With the use of external focus of attention in neuromuscular training; It has been stated that in addition to improving motor performance and biomechanical changes, the connection between the sensory areas of the brain and the thalamus has increased. It has been found to possibly reduce "noise" in the central nervous system that interferes with fine movement control and affects the outcome of movement; dopamine availability may increase, which may strengthen memory by increasing synaptogenesis processes; It has been stated in publications that newly learned motor skills can be preserved and resistance to stress and fatigue can be achieved. Considering all these situations, investigators think that young individuals with joint hypermobility may have problems with muscle strength and balance skills, which are among the physical fitness parameters. It is important to optimally evaluate physical fitness parameters in order to prevent injuries and ensure the effectiveness of the modalities used in treatment. This study was planned to investigate whether external focus of attention is effective in revealing balance skills and muscle strength at an optimal level compared to internal focus of attention in individuals with joint hypermobility.

ELIGIBILITY:
Inclusion Criteria:

* Scored 5 out of 9 or more according to Beighton scoring
* Individuals between the ages of 18-35 will be included in the research.

Exclusion Criteria:

* These individuals do not have any pathology related to the musculoskeletal system
* Those with a history of surgery within the last 6 months will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Individuals between the ages of 18-35 who score 5 or more out of 9 according to the Beighton scoring will be included in the research. Among these individuals, those with any pathology related to the musculoskeletal system or a history of surgery within the last 6 months will be excluded from the study.
  The study will be initiated with individuals who volunteer for the study as a result of the inclusion and exclusion criteria. Individuals will be evaluated for static balance, dynamic balance and lower extremity muscle strength without the use of any instructions/focus. Then, individuals' static balance, dynamic balance and lower extremity muscle strength will be evaluated according to internal and external focus techniques, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Static balance assessment: | 1-3 months
  Before starting the test, the body will be asked to position their center of gravity on the target point in as comfortable a position as possible on one leg. The dominant will be asked to stand in a single-leg stance on his legs and have his arms crossed over his shoulders. In the evaluation, participants will be asked to maintain their position on one leg with their eyes open for 20 seconds. The test will be performed 3 times and postural stability indices will be reported. Individuals will focus on their own feet while performing the internally focused static balance test. When participants switch to the externally focused test, subjects will be asked to focus on the rectangular paper placed under their feet. Additionally, individuals will be given static balance assessments without the use of any instructions/focus.
Dynamic balance assessment:Y balance test | 1-3 months
  Before starting the test, the leg lengths of the individuals will be measured from spina iliaca anterior superior (SIAS) to Medial malleolus. Then, the participants will be positioned in a standing position with one leg at the middle point of the Y-shaped platform created on the ground. Then, the patient will be asked to reach out to the directions in the test apparatus with his other extremity and touch them with his big toe. While participants focus on their own feet in the internally focused dynamic balance test, when participants switch to the externally focused test, subjects will be asked to lie down by focusing on the cone placed at the end of the test platform. The test will be performed 3 times in all directions and the averages will be recorded in cm. Additionally, individuals will receive dynamic balance assessments without the use of any instruction/focus.
Isokinetic strength evaluation | 1-3 months
  The angular values of the dynamometer and the platform on which the measurement will be made will be adjusted according to the reference values provided with the software. After the participant is placed on the platform, the overlap level of the rotation axis of the dynamometer and the anatomical axis of the knee joint will be checked. While performing the internally focused strength test, individuals will be asked to look at the quadriceps muscle previously taught by the researcher and will perform the test with this method. When the externally focused force test is started, participants will be asked to focus on the pad on the distal tibia to which subjects apply force. The total joint range of motion at which the test will be performed is determined as 0°-90°. Additionally, individuals will receive muscle strength assessments without the use of any instruction/focus.

CONTACTS AND LOCATIONS:
Overall Officials: Ali ZORLULAR, Principal Investigator — Study Principal Investigator
Locations (1):
- Rabia ZORLULAR, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smits-Engelsman B, Klerks M, Kirby A. Beighton score: a valid measure for generalized hypermobility in children. J Pediatr. 2011 Jan;158(1):119-23, 123.e1-4. doi: 10.1016/j.jpeds.2010.07.021. Epub 2010 Sep 17. PMID 20850761
- [Result] Engelbert RH, Bank RA, Sakkers RJ, Helders PJ, Beemer FA, Uiterwaal CS. Pediatric generalized joint hypermobility with and without musculoskeletal complaints: a localized or systemic disorder? Pediatrics. 2003 Mar;111(3):e248-54. doi: 10.1542/peds.111.3.e248. PMID 12612280
- [Result] Lohse KR. The influence of attention on learning and performance: pre-movement time and accuracy in an isometric force production task. Hum Mov Sci. 2012 Feb;31(1):12-25. doi: 10.1016/j.humov.2011.06.001. Epub 2011 Jul 20. PMID 21777989
- [Result] Zachry T, Wulf G, Mercer J, Bezodis N. Increased movement accuracy and reduced EMG activity as the result of adopting an external focus of attention. Brain Res Bull. 2005 Oct 30;67(4):304-9. doi: 10.1016/j.brainresbull.2005.06.035. PMID 16182938